CLINICAL TRIAL: NCT01674361
Title: A Phase II, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate Efficacy and Safety of RO4917838 in Combination With Selective Serotonin Reuptake Inhibitors in Patients With Obsessive Compulsive Disorder
Brief Title: A Study of Bitopertin (RO4917838) in Combination With Selective Serotonin Reuptake Inhibitors (SSRIs) in Participants With Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN28137
Record Dates: First submitted 2012-08-15; First posted 2012-08-28 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Bitopertin 30 mg (Experimental): Participants in Stratum 1 will receive bitopertin 30 mg from Day 1 to Week 16 in addition to their background therapy with an SSRI.
  Participants in Stratum 2 will receive placebo from Day 1 and will then start bitopertin 30 mg at the Week 2 until Week 16 in addition to their background therapy with an SSRI.
  Interventions: Drug: Bitopertin; Drug: Placebo; Drug: SSRI
- Bitopertin 10 mg (Experimental): Participants in Stratum 1 will receive bitopertin 10 mg from Day 1 to Week 16 in addition to their background therapy with an SSRI.
  Participants in Stratum 2 will receive placebo from Day 1 and will then start bitopertin 10 mg at the Week 2 until Week 16 in addition to their background therapy with an SSRI.
  Interventions: Drug: Bitopertin; Drug: Placebo; Drug: SSRI
- Placebo (Placebo Comparator): Participants (both Stratum 1 and Stratum 2) will receive placebo from Day 1 to Week 16 in addition to their background therapy with an SSRI.
  Interventions: Drug: Placebo; Drug: SSRI

INTERVENTIONS:
Drug: Bitopertin — Bitopertin once daily orally.
  Other Names: RO4917838
  Arms: Bitopertin 10 mg; Bitopertin 30 mg
Drug: Placebo — Placebo matched to bitopertin once daily orally.
Drug: SSRI — Participants will continue their background SSRI treatment as per standard of care at the same dose taken during the 8 weeks prior to Day 1. Protocol does not enforce any particular SSRI drug or regimen.

SUMMARY:
This multicenter, randomized, double-blind, parallel-group, placebo-controlled study will evaluate the efficacy and safety of bitopertin in combination with SSRI in participants with obsessive-compulsive disorder. Participants will be randomized to receive either bitopertin 30 milligrams (mg) or bitopertin 10 mg or placebo orally daily in addition to their background therapy with an SSRI. Participants will be allocated to one of two strata. Participants in Stratum 1 will start study drug on Day 1. Participants in Stratum 2 will receive placebo from Day 1 (placebo lead-in) and will then start study drug at the Week 2 visit. Participants in both strata will receive the study drug in addition to their background therapy with an SSRI until Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of OCD as per Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)
* On a stable dose of SSRI for at least 8 weeks prior to screening an between screening and Day 1
* An insufficient response to current treatment with an SSRI given at an adequate dose for at least 12 weeks prior to Day 1
* Females who are not postmenopausal or surgically sterile and who have (or may have) male sexual partners must agree to use two adequate methods of contraception as defined by protocol from the start of screening until 90 days after the last dose of study drug

Exclusion Criteria:

* Primary OCD symptom of hoarding
* More than two unsatisfactory trials within the last 2 years with different serotonin reuptake inhibitors (not including the current treatment with an SSRI) given in an adequate dose for at least 12 weeks
* Failure of more than three augmentation therapies within the last 2 years
* Undergoing acute behavioral therapy or having acute behavioral therapy that was completed less than 4 weeks prior to Day 1
* Any primary DSM-IV-TR Axis I disorder other than OCD
* Current or prior history of bipolar disorder, schizophrenia or other psychotic disorders, schizoaffective disorder, autism or autistic spectrum disorders, borderline personality disorder, or Gilles de la Tourette syndrome if symptoms have persisted into adulthood
* Any eating disorder within the last 6 months
* History of DSM-IV-TR-defined substance dependence and/or substance abuse in the last 6 months, with the exception of nicotine
* Previous treatment with bitopertin or another Glycine transporter 1 inhibitor
* Positive urine drug screening for cannabis, amphetamines (including 3,4-methylenedioxymethamphetamine [MDMA]/ecstasy), cocaine, barbiturate, and/or opiates
* Prior or current general medical condition that may impair cognition or other neuropsychiatric functioning
* Body mass index less than (<) 18.5 kilogram per square meter (kg/m^2) or greater than (>) 40 kg/m^2
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-12-31 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Total Score on Yale-Brown Obsessive Compulsive Scale (Y-BOCS) After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1), Week 12; Stratum 2: Baseline (Week 2), Week 14

SECONDARY OUTCOMES:
Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1), Week 12; Stratum 2: Baseline (Week 2), Week 14
Percentage of Participants with Response as per Pre-defined Criteria Based on the Y-BOCS and CGI | Stratum 1: Baseline (Day 1) up to Week 12; Stratum 2: Baseline (Week 2) up to Week 14
  Response will be defined as having:
  At least a 35 percent (%) reduction on the total Y-BOCS score from baseline. A much or very much improved on the Clinical Global Impression of Change (CGI-C) rating from baseline.
  A combination of at least 35% reduction on the total Y-BOCS score from baseline and much or very much improved on the CGI-C from baseline.
  Achieved remission, as shown by a total Y-BOCS score less than or equal to (≤)10.
Change From Baseline in Global Social Functioning Using Sheehan Disability Scale (SDS) Total Score After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1), Week 12; Stratum 2: Baseline (Week 2), Week 14
Change From Baseline in Global Social Functioning Using SDS Domain Scores After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1) up to Week 12; Stratum 2: Baseline (Week 2) up to Week 14
Change From Baseline in Obsessive Compulsive Inventory-Revised (OCI-R) Score After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1) up to Week 12; Stratum 2: Baseline (Week 2) up to Week 14
Change From Baseline in Columbia Suicide Severity Rating Scale After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1) up to Week 12; Stratum 2: Baseline (Week 2) up to Week 14
Change From Baseline in 36-Item Short-Form Health Survey (SF-36) - Mental Component Summary After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1) up to Week 12; Stratum 2: Baseline (Week 2) up to Week 14
Change From Baseline in SF-36 - Physical Component Summary After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1) up to Week 12; Stratum 2: Baseline (Week 2) up to Week 14
Change From Baseline in SF-36 - Domain Scores After 12 Weeks of Treatment | Stratum 1: Baseline (Day 1) up to Week 12; Stratum 2: Baseline (Week 2) up to Week 14
Area Under The Concentration-Time Curve of Bitopertin | Pre-dose (0 hour) on Day 56 (Week 8), Day 84 (Week 12), Day 98 (Week 14), Day 112 (Week 16); 3 and 6 hours post-dose on Day 112 (Week 16)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- United States (27):
  - Excell Research, Oceanside, California
  - Stanford University School of Medicine, Stanford, California
  - Yale University School of Medicine; Neuroscience Research Training Program, New Haven, Connecticut
  - Compass Research North, LLC, Leesburg, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - University of South Florida, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Carman Research, Smyrna, Georgia
  - Uni of Chicago; Centre For Advanced Medicine, Chicago, Illinois
  - Louisiana Research Associates, New Orleans, Louisiana
  - Massachusetts General Hospital - East, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Ambulatory Research Center (ARC), Department of Psychiatry, Minneapolis, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - St Louis Clinical Trials, St Louis, Missouri
  - Mount Sinai School of Medicine; Department of Psychiatry, New York, New York
  - Medical Research Network - New York, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - North Star Research, Middleburg Heights, Ohio
  - Ips Research Company, Oklahoma City, Oklahoma
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Butler Hospital - Department of Psychiatry and Human Behavior, Providence, Rhode Island
  - Clinical Neuroscience Solutions,Inc, Memphis, Tennessee
  - FutureSearch Trials, LP, Austin, Texas
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Dean Foundation, Middleton, Wisconsin
- Canada (7):
  - Chokka Center for Integrative Health, Edmonton, Alberta
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - True North Clinical Research-Halifax, Halifax, Nova Scotia
  - True North Clinical Research Kentville, Kentville, Nova Scotia
  - McMaster University - MacAnxiety Research Centre, Hamilton, Ontario
  - Sunny Johnson Medical Research Associates Inc.; Medical Research Associates, Mississauga, Ontario
  - START Clinic for Mood & Anxiety Disorders, Toronto, Ontario

REFERENCES:
- [Derived] Bandeira ID, Lins-Silva DH, Cavenaghi VB, Dorea-Bandeira I, Faria-Guimaraes D, Barouh JL, Jesus-Nunes AP, Beanes G, Souza LS, Leal GC, Sanacora G, Miguel EC, Sampaio AS, Quarantini LC. Ketamine in the Treatment of Obsessive-Compulsive Disorder: A Systematic Review. Harv Rev Psychiatry. 2022 Mar-Apr 01;30(2):135-145. doi: 10.1097/HRP.0000000000000330. PMID 35267254